CLINICAL TRIAL: NCT03489122
Title: A Randomized Control Trial Treating Depression With Yoga and Coherent Breathing Versus Walking in Veterans
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment was far from meeting target expectations, and the PO did not believe the study could achieve numbers before the end of the award
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MHBB-001-17S
Record Dates: First submitted 2018-03-28; First posted 2018-04-05 (Actual); Results first posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-04

CONDITIONS: Depressive Disorder, Major; Post Traumatic Stress Disorder
Keywords: Depressive Disorder, Major; yoga; breathing exercise; parasympathetic; anxiety; Post Traumatic Stress Disorder; polyvagal
MeSH Terms: conditions — Depressive Disorder, Major; Stress Disorders, Post-Traumatic; Anxiety Disorders | interventions — Yoga; Walking

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to a Iyengar yoga and coherent breathing or walking intervention. Two interventions a week for 12 weeks are prescribed
Who Masked: Outcomes Assessor
Masking Description: This is a behavioral intervention such that participants cannot be blinded. Participant questionnaires are fill out by participants without staff involvement. Outcome assessors: Clinicians completing the depression scales will be blinded to group assignment. Individuals analyzing magnetic resonance spectroscopy (MRS) and electrocardiogram (ECG) data will receive blinded data for analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Iyengar yoga and coherent breathing (Experimental): The yoga intervention consists of Iyengar yoga method and coherent breathing sessions for 90 minutes twice a week or a maximum of 24 interventions over the 12 week intervention.
  Interventions: Behavioral: yoga
- Walking (Active Comparator): The walking intervention consists of walking sessions at 2.5 miles an hour on a flat surface for 60 minutes twice a week or a maximum of 24 interventions over the 12 week intervention.
  Interventions: Behavioral: walking

INTERVENTIONS:
Behavioral: yoga — The yoga intervention consists of Iyengar yoga method and coherent breathing sessions for 90 minutes twice a week or a maximum of 24 interventions over the 12 week intervention.
  Arms: Iyengar yoga and coherent breathing
Behavioral: walking — The walking intervention consists of walking sessions at 2.5 miles an hour on a flat surface for 60 minutes twice a week or a maximum of 24 interventions over the 12 week intervention.
  Arms: Walking

SUMMARY:
The proposed study addresses a gap regarding the need for effective Major Depressive Disorder (MDD) treatments and the 40% of individuals treated with antidepressant medications that do not achieve full remission. This study tests a novel approach for treating MDD in a Randomized Control Trial (RTC) using yoga versus walking interventions to correct an imbalance in the Autonomic Nervous System; an over active Sympathetic Nervous System (fight or flight) an underactive Parasympathetic Nervous System (PNS) (rest, renewal and social engagement) and associated under activity in the neurotransmitter, gamma aminobutyric acid (GABA). This novel approach is complimentary to the use of antidepressant medications that primarily target the monoamine systems. Low activity in the PNS and GABA systems are also found in MDD, PTSD, and Alcohol Use Disorder, disorders representing a high healthcare burden in the Veteran population. This intervention has potential to provide relief for MDD and other disorders relevant the Veteran population

DETAILED DESCRIPTION:
Suspension of all non-essential research due to Corona Virus Disease (COVID)

Overview The study tests the hypothesis that an imbalance in the autonomic nervous system with to much sympathetic tone (Fight or Flight) and to little parasympathetic tone (rest, renewal and social engagement) and associated low activity in the neurotransmitter gamma aminobutyric acid (GABA) is associated with negative emotional states and may be a crucial underlying link between negative emotions and poor health such that the correction of these imbalances will be associated with decreased depressive symptoms in Veterans with Major Depressive Disorder (MDD). Study Design: This is a Phase 2, longitudinal, efficacy, randomized controlled trial. Veterans with MDD will be evaluated for eligibility and randomized to 12-week intervention providing two-sessions per week of either an intervention of yoga and coherent breathing at five breaths per minute or walking at 2.5 miles an hour, such that the groups are matched for metabolic demand, interaction with research staff and group effect. Depression scales will be collected at baseline and weeks 4, 8, and 12. Mood scales and RSA will be collected at baseline and pre and post interventions at weeks 4, 8, and 12. Magnetic resonance spectroscopy (MRS) data for thalamic GABA levels will be collected at baseline (Scan 1), after the 12-week intervention (Scan 2) which is immediately followed by the assigned intervention and Scan 3. The primary outcome measure is depression symptoms assessed using established rating scales. The secondary outcome measure is the thalamic GABA levels. The tertiary outcome measure is Respiratory Sinus Arrhythmia (RSA), a measure of high frequency Heart Rate Variability and a marker of parasympathetic tone. Evaluations are designed to address changes over the course of the study, and acute changes before and after interventions at week 4, 8, and 12 evaluations. Instruments: Depression scales include the Hamilton Rating Scale for Depression-17 (HDRS) and the Beck Depression Inventory II (BDI-II). Mood scales include the Spielberger State -Trait Anxiety Inventory (STAI) and the Exercise -Induced Feeling Inventory (EIFI). Post Traumatic Stress Disorder (PTSD) scales include the Clinician Administered Posttraumatic Stress Scale (CAPS) and the PTSD Check List - Civilian (PCL-C). Inclusion Criteria: The study will include 18 to 65 year old males and females Veterans with a current diagnosis of MDD who have a HDRS scores to 14 at screening. If subjects have been taking a stable dose of antidepressants that target a monoamine system for at least three months with no anticipated changes during the study, they will be allowed to continue their medication. Exclusion Criteria: The following are not allowed: history of psychosis or bipolar illness; history of suicidal ideation with intent in the last year; current mind-body practice (e.g., yoga, Tai Chi, Qigong, breathing practices, or meditation); more than three current criteria for Alcohol or Substance Use Disorder using the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) criteria; a current Substance Use Disorder, a neurologic or medical condition that could compromise subject safety or the integrity of the study. Blinding: Individuals scoring the depression scales, or analyzing the MRS and RSA data will be blind to group assignment. Hypothesis: I.a: The yoga group but not the walking group will show decreased in depressive symptoms on the HDRS and BDI-II from screening to week 12. 1.b: Subjects who are still depressed at baseline despite treatment with a stable dose (> 3 months) of antidepressants treatment will show decreased depressive symptoms in the yoga but not the walking group. 1.c: If present at baseline, there will be a greater decrease in PTSD symptoms on the CAPS in the yoga compared to the walking group. 2: There will be an increase in GABA levels over the course of the three scans in the yoga but not the walking group. 3: Over the course of the intervention and from pre to post-intervention at weeks 4, 8, and 12 there will be an improvement in the mood scales (STAI and EIFI), and increase in RSA in the yoga but not the walking group.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English
* Understands the risks and benefits of the study as listed in the Post Consent Quiz
* Females must agree to use an acceptable form of birth control [Human Subjects]
* Females are not pregnant and do not intend to become pregnant during the study
* Meets criteria for MDD on the Mini-International Neuropsychiatric Interview (MINI)
* Hamilton Rating Scale for Depression (HDRS) scores to 14 at screening
* If subjects have been taking antidepressants that target a monoamine system, the dose has been stable for at least three months with no anticipated changes during the study
* If subjects have been in a stable form of psychotherapy for three months, with no anticipated changes in their psychotherapy during the study (this would exclude time-limited manual-driven therapies such Cognitive Behavioral Therapy)
* Reliable contact information provided
* Has completed all required screening instruments and evaluations

Exclusion Criteria:

* History of psychosis
* History of bipolar illness
* History of suicidal ideation with intent and or a suicide attempt in the last year
* Desire to be treated for MDD with a new treatment during the study such as pharmacotherapy, somatic therapy or psychotherapy
* Current mind-body practice defined as more than 6 one-hour sessions in the last 6 months

  * yoga
  * Tai Chi
  * Qigong
  * breathing practices, or meditation
* Participates in physical exercise > 5 hours/week that is equivalent to or greater than 6 metabolic equivalents (METs) in intensity
* Has been treated psychotropic medications such as mood stabilizers

  * Valproic Acid
  * Carbamazepine
  * Lithium
* Benzodiazepines or pain medication other than Non Steroidal Anti-Inflammatory Drugs (NSAIDS) in the last three months except for procedure related pain management

  * dental procedures
* Has more than three current criteria for Alcohol or Substance Use Disorder using DSM-V criteria
* Has a neurologic or medical condition that in the opinion of the PI could compromise subject safety or the integrity of the study
* In the opinion of the PI, would not be expected to complete the study, or their participation would be jeopardized subject safety or the integrity of the study
* Has an Axis-I diagnosis, other than depression except as listed, that in the opinion of the PI would interfere with the subject's participation in this study
* Anxiety disorders with current symptoms that would impair participation in the study

  * Obsessive Compulsive Disorder (OCD) or agoraphobia that would prevent intervention attendance
  * Post Traumatic Stress Disorder with dissociation or flashbacks that could be triggered by the yoga intervention
  * Claustrophobia that would prevent scanning
* Traumatic Brain Injury (TBI) with greater than 30 minutes loss of consciousness
* Must have a period of 48 hours of no alcohol use and 24 hours of no nicotine use on the Timeline Followback (TLFB) to participate in scanning given the effects of tobacco smoke and alcohol consumption on the GABA system

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris C Streeter, MD, Principal Investigator — VA Bedford HealthCare System, Bedford, MA
Locations (1):
- VA Bedford HealthCare System, Bedford, MA, Bedford, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Mechanisms for public access to final data sets underlying publications from this research: A limited Dataset (LDS) will be created and shard pursuant to a Data Use Agreement (DUA) appropriately limiting use of the dataset and prohibiting the recipient form identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the data set.
Time Frame: Final data sets will be available electronically after publication of the hypotheses or 5 years after protocol completion.
Access Criteria: Data will be provided to qualified researchers after the written request of their data use plan is approved in writing by the Bedford VA research office. Original research team members are allowed to review potential publications to assure final data set use is consistent with collection circumstances. Member that review potential publications will be included as authors.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Iyengar Yoga and Coherent Breathing | Walking
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: study was terminated due to extremely low enrollment
Groups:
- Total: Total of all reporting groups
Arm/Group | Iyengar Yoga and Coherent Breathing | Walking | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 39 [39 to 39] | 54 [54 to 54] | 46.5 [39 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 1 | 2
Hamilton Depression Rating Scales [Mean (Full Range); unit: units on a scale] — 17-item clinician administered scale. The maximum score being 52. Scores of 0-7 are considered as being normal, 8-16 suggest mild depression, 17-23 moderate depression and scores over 24 are indicative of severe depression.
  units on a scale | 26 [26 to 26] | 17 [17 to 17] | 21.5 [17 to 26]

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scales Change
Description: The Hamilton Depression Rating Scale for Depression is a clinician administered scale used to assess depressive symptoms. A 17-item clinician administered scale. The maximum score being 52. Scores of 0-7 are considered as being normal, 8-16 suggest mild depression, 17-23 moderate depression and scores over 24 are indicative of severe depression. A score of 0-7 is generally accepted to be within the normal), while a score of 20 or higher (indicating at least moderate severity) is usually required for entry into a clinical trial.
Time Frame: Screening, week 4, week 8, week 12
Population: subject was lost to follow up
Measure: Number; unit: units on a scale
Arm/Group | Iyengar Yoga and Coherent Breathing | Walking
Number analyzed (Participants) | 1 | 1
units on a scale
  Screening | 27 | 17
  Week 4 | 16 | 5
  Week 8: number analyzed (Participants) | 1 | 0
  Week 8 | 13 |
  Week 12: number analyzed (Participants) | 1 | 0
  Week 12 | 16 |

2. Secondary Outcome: Gamma Amino Butyric Acid (GABA) Change
Description: Magnetic Resonance Spectroscopy (MRS) will be used to measure GAB levels in the left thalamus Scan 1 prior to randomization, Scan 2 after the 12-week intervention, immediately after Scan 2 there will be a yoga or walking intervention determined by group assignment that will be immediately followed by Scan 3.
  Participation in the study maybe up to 22 weeks due to the need to scan females who are cycling in the first half of their menstrual cycle.
Time Frame: 12 weeks, up to 22 weeks
Population: Although a contract was in place, no scans were ever performed on the participants and therefore, data were never collected. Additional details regarding why, specifically, scans were ultimately not performed were not provided by the PI who has retired.
Arm/Group | Iyengar Yoga and Coherent Breathing | Walking
Number analyzed (Participants) | 0 | 0

3. Other Pre Specified Outcome: Respiratory Sinus Arrhythmia (RSA)
Description: Electrocardiogram data will be obtained at rest, during a 3 minute aerobic step test and during recovery for RSA analysis at the above times. RSA measures the vagal component of heart rate variability. It is a marker of parasympathetic activity.
Time Frame: Before Scans 1-3, before and after the week 4, 8, and 12 evaluations
Population: this data was not collected
Arm/Group | Iyengar Yoga and Coherent Breathing | Walking
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Clinician Administered Posttraumatic Stress Scale (CAPS)
Description: This is an exploratory measure. Clinician Administered Posttraumatic Stress Scale (CAPS) is a clinician administered interview to diagnose the severity of Post Traumatic Stress Disorder (PTSD). Decreasing CAPS scores are a marker of decreasing PTSD symptoms. CAPS scores of greater than or equal to 20 indicate at least mild PTSD.
Time Frame: Screening and week 12 evaluation
Population: this data was not collected
Arm/Group | Iyengar Yoga and Coherent Breathing | Walking
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: State Trait Anxiety Inventory-State (STAI)
Description: The State-Trait Anxiety Inventory (STAI) is a self-administered instrument designed for serial assessment of state anxiety. It has 20 items and is rated on a 4-point scale. Responses for the scale assess intensity of current feelings "at this moment": 1) not at all, 2) somewhat, 3) moderately so, and 4) very much so. The range of scores is 20-80 with higher scores indicating higher anxiety.
Time Frame: Screening, and pre and post the week 4, 8, and 12 evaluations
Population: subject was lost to follow up
Measure: Number; unit: units on a scale
Arm/Group | Iyengar Yoga and Coherent Breathing | Walking
Number analyzed (Participants) | 1 | 1
units on a scale
  Screening | 46 | 40
  Pre-Week 4 | 40 | 43
  Post-Week 4 | 36 | 32
  Pre-Week 8: number analyzed (Participants) | 1 | 0
  Pre-Week 8 | 44 |
  Post-Week 8: number analyzed (Participants) | 1 | 0
  Post-Week 8 | 41 |
  Pre-Week 12: number analyzed (Participants) | 1 | 0
  Pre-Week 12 | 37 |
  Post-Week 12: number analyzed (Participants) | 1 | 0
  Post-Week 12 | 45 |

6. Other Pre Specified Outcome: Exercise Induced Feeling Inventory (EIFI)
Description: Exercise-Induced Feeling Inventory (EIFI) is a self-administered instrument designed to assess four distinct feeling states associated with bouts of physical activity. It consists of 12 items that capture 4 distinct feeling states: Revitalization, Tranquility, Positive Engagement, and Physical Exhaustion. Improvements are associated with increased scores on Revitalization, Tranquility, Positive Engagement, and decreased scores on Physical Exhaustion. All items are scored on a 5-point scale anchored from 0 (do not feel) to 4 (feel very strongly). The range of scores is 0-48 with higher scores on the EFI total and subscales indicate more positive mood states, except on the Physical Exhaustion subscale where high scores indicate greater physical exhaustion.
Time Frame: Screening, and pre and post the week 4, 8, and 12 evaluations
Population: subject was lost to follow up
Measure: Number; unit: units on a scale
Arm/Group | Iyengar Yoga and Coherent Breathing | Walking
Number analyzed (Participants) | 1 | 1
units on a scale
  Screening | 19 | 16
  Pre-Week 4 | 12 | 10
  Post-Week 4 | 13 | 13
  Pre-Week 8: number analyzed (Participants) | 1 | 0
  Pre-Week 8 | 22 |
  Post-Week 8: number analyzed (Participants) | 1 | 0
  Post-Week 8 | 25 |
  Pre-Week 12: number analyzed (Participants) | 1 | 0
  Pre-Week 12 | 17 |
  Post-Week 12: number analyzed (Participants) | 1 | 0
  Post-Week 12 | 19 |

7. Other Pre Specified Outcome: Pittsburgh Sleep Quality Inventory
Description: The Pittsburgh Sleep Quality Index (PSQI) is a self-reported questionnaire which assesses sleep quality and disturbances over a 1-month time interval. The PSQI consists of 24 questions or items measuring seven dimensions from 0 (best) to 3 (worst): subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score from 0 to 21, with 0-4 indicating "good" sleep and 5-21 indicating "poor" sleep.
Time Frame: Obtained at screening, and weeks 4, 8, and 12 evaluations.
Population: subject was lost to follow up
Measure: Number; unit: units on a scale
Arm/Group | Iyengar Yoga and Coherent Breathing | Walking
Number analyzed (Participants) | 1 | 1
units on a scale
  Screening | 14 | 14
  Week 4 | 7 | 6
  Week 8: number analyzed (Participants) | 1 | 0
  Week 8 | 8 |
  Week 12: number analyzed (Participants) | 1 | 0
  Week 12 | 7 |

8. Other Pre Specified Outcome: Beck Depression Inventory II (BDI-II)
Description: Beck Depression Inventory (BDI-II) is a 21-item self-administered instrument designed for the assessment of depressive symptoms, with higher scores reflecting greater severity. The items are scored on a 4-point scale where answers are assigned a point value from zero to three. Minimal Depression: Zero - 13; Mild Depression: 14 - 19; Moderate Depression: 20 - 28; Severe Depression: 29 - 63
Time Frame: Screening, weeks 4, 8, 12 evaluations
Population: subject was lost to follow up
Measure: Number; unit: units on a scale
Arm/Group | Iyengar Yoga and Coherent Breathing | Walking
Number analyzed (Participants) | 1 | 1
units on a scale
  Screening | 31 | 25
  Week 4 | 25 | 16
  Week 8: number analyzed (Participants) | 1 | 0
  Week 8 | 35 |
  Week 12: number analyzed (Participants) | 1 | 0
  Week 12 | 32 |

9. Other Pre Specified Outcome: Post Traumatic Check List - Civilian (PCL)
Description: PTSD Check List - Civilian (PCL-5) is a 20-item self-administered scale and is rated on a 5-point scale (0="Not at all" to 4= "Extremely") corresponding to Diagnostic and Statistical Manual of Mental Disorders (DSM) IV criteria for PTSD. Because not all Veterans have combat experience and not all trauma is from a military experience, the civilian version of the PCL will be used. A total symptom severity score (range - 0-80) is obtained by summing the scores for each of the 20 items
Time Frame: Screening, and weeks 4, 8, 12 evaluations
Population: subject was lost to follow up
Measure: Number; unit: units on a scale
Arm/Group | Iyengar Yoga and Coherent Breathing | Walking
Number analyzed (Participants) | 1 | 1
units on a scale
  Screening | 44 | 43
  Week 4 | 41 | 36
  Week 8: number analyzed (Participants) | 1 | 0
  Week 8 | 57 |
  Week 12: number analyzed (Participants) | 1 | 0
  Week 12 | 55 |

10. Other Pre Specified Outcome: Brief Pain Inventory (BPI)
Description: Brief Pain Inventory (BPI) consists of 9 items rated on an eleven point Likert Scale of pain intensity (0-10) will be used to assess pain over the last 24 hours. The range of scores is 0-90 with higher total scores indicate greater severity and impact of pain.
Time Frame: Weeks 4, 8, 12 evaluations.
Population: subject was lost to follow up
Measure: Number; unit: units on a scale
Arm/Group | Iyengar Yoga and Coherent Breathing | Walking
Number analyzed (Participants) | 1 | 1
units on a scale
  Week 4 | 42 | 0
  Week 8: number analyzed (Participants) | 1 | 0
  Week 8 | 51 |
  Week 12: number analyzed (Participants) | 1 | 0
  Week 12 | 49 |

ADVERSE EVENTS:
Time Frame: While participants were to be screened weekly for Adverse Events (to include the 12-week intervention and follow-up calls at 2 and 6 months post-intervention) they were actually monitored/assessed for a shorter duration of time. The participant in the yoga arm was followed weekly throughout the 12-week intervention, and the participant in the walking arm was followed weekly for 7 weeks until lost to follow-up due to their personal scheduling constraints.
Arm/Group | Iyengar Yoga and Coherent Breathing | Walking
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

LIMITATIONS AND CAVEATS:
COVID forced the study to have virtual interventions which affected enrollment. Early termination leading to only one participant per study arm prevented analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-03-07): https://cdn.clinicaltrials.gov/large-docs/22/NCT03489122/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-20): https://cdn.clinicaltrials.gov/large-docs/22/NCT03489122/SAP_001.pdf